CLINICAL TRIAL: NCT00846625
Title: Study of Uveitic Macular Edema Treated With Ranibizumab or Steroids Following a Periocular Steroid Injections in Patients on Steroid Sparing Agents or Low Dose Steroids
Brief Title: Study of Uveitic Macular Edema Treated With Ranibizumab or Steroids
Acronym: SURFING
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient enrollment (no subjects were enrolled)
Sponsor: University of Utah (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Albert T. Vitale, MD, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 34035
Record Dates: First submitted 2009-02-18; First posted 2009-02-19 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Macular Edema; Uveitis
Keywords: Biomedical research; Macular Edema; Uveitis; Ranibizumab; Steroids
MeSH Terms: conditions — Macular Edema; Uveitis | interventions — Triamcinolone; Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Ranibizumab (0.5 mg)
  Interventions: Drug: ranibizumab
- 2 (Active Comparator): Triamcinolone (4 mg/0.1 ml)
  Interventions: Drug: triamcinolone

INTERVENTIONS:
Drug: triamcinolone — Intravitreal injection (4 mg/0.1 ml)
  Other Names: Triescence
  Arms: 2
Drug: ranibizumab — Intravitreal injection, 0.5 mg
  Other Names: Lucentis
  Arms: 1

SUMMARY:
This is a pilot study to investigate the safety and efficacy of intravitreally administered ranibizumab (Lucentis) compared to steroid injection for the treatment of macular edema due to chronic non-infectious uveitis. There is currently no FDA-approved therapy for this condition, however intravitreal injection of corticosteroids, in conjunction with oral steroids and/or immunomodulatory drug agents, has become the mainstay of therapy. Ranibizumab is a recombinant monoclonal antibody antigen-binding fragment that neutralizes the active forms of vascular endothelial growth factor (VEGF), which is believed to contribute to the etiology of inflammation and neovascularization. Ranibizumab is FDA-approved for the treatment of neovascular age-related macular degeneration.

DETAILED DESCRIPTION:
This is a proof of concept study to assess the safety and potential efficacy of ranibizumab in this patient population. Since it is common clinical practice to perform regional periocular injections of steroids in patients with uveitic macular edema, only patients who are refractory to periocular steroids will be enrolled in the study. The 0.5 mg dose of ranibizumab will be given intravitreally since this dose and route has been found to be safe and efficacious in prior studies. A dosing regimen has not been established for ranibizumab in patients with uveitis, so patients will be assessed and treated monthly as needed. Triamcinolone 4mg intravitreal injection will be the steroid treatment, and patients will also be assessed monthly and retreated every three months as needed.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* History of non-infectious uveitis w chronic cystoid macular edema
* Refractory to therapy w periocular steroids; Last periocular steroid injection a minimum of 3 months prior to study enrollment
* Currently using oral steroids (< or = 10 mg/day) and/or steroid sparing agents
* BCVA between 20/40 and 20/400
* IOP between 5 mmHg and 30 mmHg
* Media clarity sufficient for OCT measurement

Exclusion Criteria:

* Women known to be pregnant or have a positive urine pregnancy test; Pre-menopausal women not using adequate contraception during the study
* Prior treatment for CME with Macugen or Avastin in the study eye
* History of stroke
* Presence of vitreous hemorrhage or epiretinal membrane in the study eye
* Active infectious conjunctivitis, keratitis, scleritis or endophthalmitis in either eye
* Presence or history of uncontrolled glaucoma
* Known allergy or hypersensitivity to any component of the study drug
* Major surgery planned during the next 6 months
* Simultaneous participation in another clinical investigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-11; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Ocular adverse events | 12 months

SECONDARY OUTCOMES:
Resolution of macular edema by OCT measurement | 3, 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Albert T Vitale, MD, Principal Investigator — University of Utah
Locations (1):
- John Moran Eye Center, Salt Lake City, Utah, United States